CLINICAL TRIAL: NCT05152147
Title: A Randomized, Multicenter, Phase 3 Study of Zanidatamab in Combination With Chemotherapy With or Without Tislelizumab in Subjects With HER2-positive Unresectable Locally Advanced or Metastatic Gastroesophageal Adenocarcinoma (GEA)
Brief Title: A Study of Zanidatamab in Combination With Chemotherapy Plus or Minus Tislelizumab in Patients With HER2-positive Advanced or Metastatic Gastric and Esophageal Cancers
Acronym: HERIZON-GEA-01
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: BeOne Medicines LTD (Unknown); BeOne Pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZWI-ZW25-301; 2021-000296-36 (EudraCT Number); jRCT2061230026 (Registry Identifier: Japan Registry for Clinical Trials (jRCT)); 2023-510319-20-00 (EU CTIS Number)
Expanded Access: NCT04578444 (No longer available)
Record Dates: First submitted 2021-11-05; First posted 2021-12-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Gastric Neoplasms; Gastroesophageal Adenocarcinoma; Esophageal Adenocarcinoma
Keywords: HER2; Bispecific antibody; Biparatopic antibody; Immunotherapy; Gastric cancers; Esophageal cancers; Chemotherapy; FP; Capecitabine; Cisplatin; 5-FU; Oxaliplatin; Gastroesophageal adenocarcinoma; CAPOX; Programmed cell death receptor 1 (PD-1); Anti-PD-1; Anti PD-1; JZP598
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — zanidatamab; tislelizumab; Trastuzumab; Capecitabine; Oxaliplatin; Cisplatin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: multi-cohort, open-label, multicenter study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Active Comparator): Trastuzumab (Herceptin®) plus physician's choice of capecitabine plus oxaliplatin (CAPOX) or 5-fluorouracil (5-FU) plus cisplatin (FP)
  Interventions: Drug: Trastuzumab; Drug: Capecitabine; Drug: Oxaliplatin; Drug: Cisplatin; Drug: 5-Fluorouracil
- Arm B (Experimental): Zanidatamab plus physician's choice of CAPOX or FP
  Interventions: Drug: Zanidatamab; Drug: Capecitabine; Drug: Oxaliplatin; Drug: Cisplatin; Drug: 5-Fluorouracil
- Arm C (Experimental): Zanidatamab and tislelizumab plus physician's choice of CAPOX or FP
  Interventions: Drug: Zanidatamab; Drug: Tislelizumab; Drug: Capecitabine; Drug: Oxaliplatin; Drug: Cisplatin; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Zanidatamab — Administered IV
  Other Names: ZW25; JZP598; ZIIHERA®
  Arms: Arm B; Arm C
Drug: Tislelizumab — Administered IV
  Arms: Arm C
Drug: Trastuzumab — Administered intravenously (IV)
  Other Names: Herceptin®
  Arms: Arm A
Drug: Capecitabine — Administered orally (PO bid)
Drug: Oxaliplatin — Administered IV
Drug: Cisplatin — Administered IV
Drug: 5-Fluorouracil — Administered IV

SUMMARY:
This study is being done to find out if zanidatamab, when given with chemotherapy plus or minus tislelizumab, is safe and works better than trastuzumab given with chemotherapy.

The patients in this study will have advanced human epidermal growth factor 2 (HER2)-positive stomach and esophageal cancers that are no longer treatable with surgery (unresectable) or chemoradiation, and/or have grown or spread to other parts of the body (metastatic).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable locally advanced, recurrent or metastatic HER2-positive gastroesophageal adenocarcinoma (adenocarcinomas of the stomach or esophagus, including the gastroesophageal junction), defined as 3+ HER2 expression by IHC or 2+ HER2 expression by IHC with ISH positivity per central assessment. Subjects with esophageal adenocarcinoma must not be eligible for combined chemoradiotherapy at the time of enrollment
* Assessable (measurable or non-measurable) disease as defined by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1, assessed within 3 days prior to randomization
* Adequate organ function
* Left ventricular ejection fraction (LVEF) ≥ 50% as determined by either echocardiogram or multiple gated acquisition scan (MUGA)

Exclusion Criteria:

* Prior treatment with a HER2-targeted agent, with the exception of subjects who received HER2-targeted treatment for breast cancer > 5 years prior to initial diagnosis of GEA
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2 or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Prior treatment with systemic antineoplastic therapy or intraperitoneal chemotherapy for unresectable locally advanced, recurrent or metastatic GEA
* Untreated central nervous system (CNS) metastases, symptomatic CNS metastases, or radiation treatment for CNS metastases within 4 weeks prior to randomization. Stable, treated brain metastases are allowed (defined as subjects who are completely off steroids and anticonvulsants and are neurologically stable with no evidence of radiographic progression for at least 4 weeks prior to randomization)
* Known history of or ongoing leptomeningeal disease (LMD)
* Known additional malignancy that is not considered cured or that has required treatment within the past 3 years
* Known active hepatitis
* Any history of human immunodeficiency virus (HIV) infection
* Known SARS-CoV-2 infection; subjects with prior infection that has resolved per local institutions' requirements and screening guidance are eligible
* QTc Fridericia (QTcF) > 470 ms
* Clinically significant cardiac disease, such as ventricular arrhythmia requiring therapy, uncontrolled hypertension or any history of symptomatic congestive heart failure (CHF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 920 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) by BICR | Up to 2.5 years
  The time from randomization to the date of documented disease progression (per Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1) as assessed by blinded independent central review (BICR) or death from any cause
Overall survival | Up to 3.5 years
  The time from randomization to death due to any cause

SECONDARY OUTCOMES:
Confirmed objective response rate (ORR) by BICR | Up to 2.5 years
  Number of patients who achieved a best overall response of complete response (CR) or (PR) as determined per RECIST 1.1 as assessed by BICR
Duration of response (DOR) by BICR | Up to 2.5 years
  The time from the first objective response (CR or PR) per BICR to documented progressive disease per RECIST 1.1 as assessed by BICR or death from any cause
PFS per Investigator assessment | Up to 2.5 years
  The time from randomization to the date of documented disease progression (per RECIST 1.1) as assessed by Investigator or death from any cause
Confirmed ORR per Investigator assessment | Up to 2.5 years
  Number of patients who achieved a best overall response of CR or PR as determined per RECIST 1.1 as assessed by Investigator
DOR per Investigator assessment | Up to 2.5 years
  The time from the first objective response (CR or PR) per Investigator to documented progressive disease per RECIST 1.1 as assessed by Investigator or death from any cause
Assessment of Contribution of Components based on Progression-free Survival (PFS) by BICR | Up to 2.5 years
  The time from randomization to the date of documented disease progression (per Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1) as assessed by blinded independent central review (BICR) or death from any cause
Assessment of Contribution of Components based on Overall Survival | Up to 3.5 years
  The time from randomization to death due to any cause
Incidence of adverse events | Up to 2 years
  Number of subjects who experienced adverse events or serious adverse events
Incidence of clinical laboratory abnormalities | Up to 2 years
  Number of patients who experienced a maximum severity of Grade 3 or higher post-baseline laboratory abnormality, including either hematology or chemistry. Grades are defined using National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 5.0
Health-related quality of life (HRQoL) as assessed by the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (core cancer questionnaire) C30 (QLQ-C30) | Up to 2.5 years
  Changes from baseline in the EORTC QLQ-C30 scores
HRQoL as assessed by the EORTC Quality of Life Questionnaire (oesophago-gastric module) OG25 (QLQ-OG25) | Up to 2.5 years
  Changes from baseline in the EORTC QLQ-OG25 scores
HRQoL as assessed by the EuroQol 5-dimensions 5-levels (EQ-5D-5L) questionnaire | Up to 2.5 years
  Changes from baseline in the EORTC EQ-5D-5L questionnaire scores
Serum concentration of zanidatamab and tislelizumab | Up to 2 years
Incidence of anti-drug antibodies (ADAs) | Up to 2 years
  Number of patients who develop ADAs

CONTACTS AND LOCATIONS:
Locations (226):
- Argentina (7):
  - Hospital de Gastroenterología Dr Bonorino Udaondo, Buenos Aires
  - Instituto de Investigaciones Metabólicas - IDIM, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Fundación Centro de Medicina Nuclear y Molecular ER, Córdoba
  - Centro Médico Privado CEMAIC, Córdoba
  - Centro de Investigación Pergamino S.A., Pergamino
  - Centro de Investigación Clínica - Clínica Viedma, Viedma
- Australia (4):
  - Flinders Medical Centre, Bedford Park
  - Austin Health, Heidelberg
  - Liverpool Hospital, Liverpool
  - Fiona Stanley Hospital, Murdoch
- Belgium (5):
  - Imelda VZW, Bonheiden
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
- Brazil (11):
  - Centro Integrado de Pesquisa - CIP, Barretos
  - Fundação Pio XII Hospital de Câncer de Barretos, Barretos
  - Cenantron - Centro Avancado de Tratamento Oncologico Ltda, Belo Horizonte
  - Centro de Pesquisas Clínicas/Fundação Doutor Amaral Carvalho, Brasília
  - Instituto Do Câncer Do Ceará ICC, Fortaleza
  - Hospital de Clinicas de Porto Alegre (HCPA) - PPDS, Porto Alegre
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital Nossa Senhora Da Conceição, Porto Alegre
  - Núcleo de Pesquisa Clínica da Rede São Camilo, Santo André
  - Instituto do Cancer do Estado de São Paulo ICESP, São Paulo
  - Instituto de Oncologia de Sorocaba, Sorocaba
- Princess Margaret Cancer Centre, Toronto, Canada
- Chile (7):
  - Centro Internacional de Estudios Clinicos CIEC, Santiago, Region Metropolitan
  - Fundación Arturo López Pérez (FALP) - PPDS, Providencia, Santiago Metropolitan
  - Centro de Estudios Clínicos SAGA SpA, Providencia
  - Sociedad Oncovida S.A, Santiago
  - Icegclinic, Santiago
  - BIOCINETIC SpA, Santiago
  - Sociedad de Investigaciones Medicas Limitada, Temuco
- China (51):
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Beijing Cancer Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Luhe Hospital, Capital Medical University, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Hunan Cancer Hospital, Changsha
  - Changzhi People's Hospital, Changzhi
  - Changzhou First People's Hospital, Changzhou
  - Sichuan Cancer Hospital & Institute, Chengdu
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Fujian Cancer Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - Hainan General Hospital, Haikou
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou
  - Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Provincial Cancer Hospital, Hefei
  - The Second Affiliated Hospital of Anhui Medical University, Hefei
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - Shandong Cancer Hospital, Jinan
  - Jinan Central Hospital, Jinan
  - Yunnan Cancer Hospital, Kunming
  - The First Hospital of Lanzhou University, Lanzhou
  - Gansu Cancer Hospital, Lanzhou
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital ,The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Ruijin hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - Fudan University Affiliated Zhongshan Hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai General Hospital, Shanghai
  - Liaoning Cancer Hospital & Institute, Shenyang
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin Medical University General Hospital, Tianjin
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - The Tonghua Central Hospital, Tonghua
  - Cancer Hospital affiliated to Xinjiang Medical University, Ürümqi
  - Weihai Municipal Hospital, Weihai
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Union Hospital Tongji Medical College HuaZhong University of Science and Technology, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - Affiliated Hospital of Jiangnan University, Wuxi
  - First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Northern Jiangsu People's Hospital, Yangzhou
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- North Estonia Medical Centre Foundation, Tallinn, Estonia
- France (12):
  - CHU de Bordeaux - Hopital Haut Leveque, Pessac, Gironde
  - Sainte-Catherine, Institut du Cancer Avignon Provence, Avignon
  - EDOG - Institut Bergonie - PPDS, Bordeaux
  - Universite de Bourgogne - Faculte de Medecine - IN, Dijon
  - Centre Hospitalier Universitaire Grenoble Alpes - Hopital Albert Michallon, Grenoble
  - Centre Léon Berard, Lyon
  - EDOG Institut de Cancerologie de l'Ouest - PPDS, Nantes
  - CHRU de Poitiers La Miletrie, Poitiers
  - EDOG - Centre Eugene Marquis Centre Regional de Lutte Contre Le Cancer - PPDS, Rennes
  - CHRU de Brest - Hopital Morvan, Saint-Priest-en-Jarez
  - Hôpital de Rangueil, Toulouse
  - Hôpital Saint Antoine, Villejuif
- Georgia (2):
  - Research Institute of Clinical Medicine, Tbilisi
  - High Technology Hospital MedCenter Ltd, Tbilisi
- Institut für Klinisch-Onkologische Forschung, Frankfurt am Main, Hesse, Germany
- Greece (4):
  - Attikon University General Hospital, Athens
  - Bioclinic Thessaloniki Oncology Department, Thessaloniki
  - Agios Loucas Clinic SA, Thessaloniki
  - Interbalkan Medical Center of Thessaloniki Oncology Department, Thessaloniki
- Guatemala (3):
  - Clinica Medica Especializada CELAN, Guatemala City
  - Grupo Medico Angeles, Guatemala City
  - Centro Medico Integral de Cancerologia CEMIC, Salcajá
- India (6):
  - All India Institute of Medical Sciences, Bhubaneswar, Bhubaneswar
  - Artemis Hospital, Gūrgaon
  - MNJ Institute of Oncology and Regional Cancer Centre, Hyderabad
  - Indraprastha Apollo Hospitals, New Delhi
  - Regional Cancer Centre Indira Gandhi Institute of Medical Sciences, Patna
  - HCG City Cancer Center, Vijayawada
- St James's Hospital, Dublin, Ireland
- Italy (12):
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi, Bologna
  - Fondazione del Piemonte per l'Oncologia (IRCCS), Candiolo
  - Ospedale Policlinico San Martino, Genova
  - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori IRST - PPDS, Meldola
  - Ospedale San Raffaele S.r.l. - PPDS, Milan
  - Istituto Nazionale Dei Tumori, Milan
  - ASST Grande Ospedale Metropolitano Niguarda - Presidio Ospedaliero Ospedale Niguarda, Milan
  - Azienda Ospedaliero Universitaria Di Modena Policlinico, Modena
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Fondazione Policlinico Universitario A Gemelli, Rome
  - Centro Ricerche Cliniche Di Verona, Verona
  - Azienda ULSS 8 "Berica" - Ospedale San Bortolo, Vicenza
- Japan (22):
  - Chiba Cancer Center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Gifu University Hospital, Gifu, Gihu
  - Gunma Prefectural Cancer Center, Ota-shi, Gunma
  - Hyogo Cancer Center, Akashi-shi, Hyôgo
  - Ibaraki Prefectural Central Hospital, Kasama-Shi, Ibaraki
  - Kagawa University Hospital, Kita-Gun Miki-Cho, Kagawa-ken
  - Kanagawa Cancer Center, Yokohama-Shi Asahi-Ku, Kanagawa
  - Kumamoto University Hospital - Honjo-Kuhonji Campus A, Chuo-Ku, Kumamoto
  - Kyoto University Hospital, Sakyo-ku, Kyoto-shi
  - Osaki Citizen Hospital, Osaki-Shi, Miyagi
  - Kurashiki Central Hospital, Kurashiki-Shi, Okayama-ken
  - Osaka University Hospital, Suita-Shi, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki-Shi, Osaka
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - National Cancer Center Hospital, Chūōku
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Saitama Cancer Center, Ina
  - Shikoku Cancer Center, Matsuyama
  - Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Ōsaka-sayama
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Tokyo
- Malaysia (3):
  - Hospital Pulau Pinang, George Town
  - Sarawak General Hospital, Kuching
  - National Cancer Institute ( Institut Kanser Negara), Putrajaya
- Mexico (3):
  - Health Pharma Professional Research S.A de C.V., Mexico City
  - Hospital Universitario Dr. Jose Eleuterio González, Monterrey
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
- Netherlands (3):
  - Catharina Hospital, Eindhoven
  - Leids Universitair Medisch Centrum, Leiden
  - ETZ-Elisabeth, Tilburg
- Poland (2):
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz
  - Centrum Onkologii Instytut im. Marii Sklodowskiej-Curie, Warsaw
- Portugal (7):
  - Hospital Garcia de Orta, Almada
  - Centro Hospitalar E Universitário de Coimbra EPE, Coimbra
  - Hospital Senhora da Oliveira - Guimaraes, E.P.E, Guimarães
  - Centro Hospitalar Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Unidade Local de Saúde de Matosinhos SA, Matosinhos Municipality
  - Centro Hospitalar do Porto EPE, Porto
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe - PPDS, Porto
- Romania (4):
  - Fundeni Clinical Institute, Bucharest
  - Prof Dr I Chiricuta Institute of Oncology - PPDS, Cluj-Napoca
  - Medisprof SRL, Cluj-Napoca
  - Oncology Center Sfantul Nectarie, Craiova
- Serbia (4):
  - University Clinical Center of Serbia - PPDS, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
  - University Clinical Center Nis, Niš
- National Cancer Center Singapore, Singapore, Singapore
- Wilgers Oncology Centre, Pretoria, South Africa
- South Korea (16):
  - Hallym University Sacred Heart Hospital, Anyang-si
  - Dong-A University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Gachon University Gil Medical Center, Incheon
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (13):
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Institut Català d'Oncologia (Hospital Duran y Reynals), L'Hospitalet de Llobregat
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Regional Universitario de Malaga - Hospital General, Málaga
  - Complejo Asistencial Universitario de Salamanca - H. Clinico, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
- Thailand (2):
  - Songklanagarind Hospital, Hat Yai
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
- Turkey (Türkiye) (6):
  - Hacettepe Universitesi Kanser Enstitusu, Ankara
  - Trakya University Medical Faculty, Edirne
  - Dokuz Eylul Universitesi, Izmir
  - Acibadem Adana Hospital, Seyhan
  - Medical Park Trabzon Yildizli, Trabzon
  - Dr. Abdurrahman Yurtaslan Ankara Onkology Training and Research Hospital, Yenimahalle
- The Municipal Enterprise Volyn Regional Medical Oncology Centre of the Volyn Regional Council, Lutsk, Ukraine
- United Kingdom (8):
  - Bristol Haematology and Oncology Centre, Bristol
  - Western General Hospital Edinburgh - PPDS, Edinburgh
  - St James University Hospital, Leeds
  - Guy's and St Thomas' NHS Foundation Trust - Guy's Hospital, London
  - Royal Marsden Hospital - London, London
  - Royal Marsden Hospital - Surrey, London
  - Edith Cavell Hospital, Peterborough
  - Weston Park Cancer Centre, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee KW, Bai LY, Jung M, Ying J, Im YH, Oh DY, Cho JY, Oh SC, Chao Y, Kim JW, Chen Y, Li V, Chen S, Kang YK. Phase Ib/II Study of Zanidatamab in Combination with Tislelizumab and Chemotherapy in First-Line HER2-Positive Gastric/Gastroesophageal Junction Adenocarcinoma. Clin Cancer Res. 2026 Jan 16;32(2):312-323. doi: 10.1158/1078-0432.CCR-24-4295. PMID 41324998
- [Derived] Tabernero J, Shen L, Elimova E, Ku G, Liu T, Shitara K, Lin X, Boyken L, Li H, Grim J, Ajani J. HERIZON-GEA-01: Zanidatamab + chemo +/- tislelizumab for 1L treatment of HER2-positive gastroesophageal adenocarcinoma. Future Oncol. 2022 Sep;18(29):3255-3266. doi: 10.2217/fon-2022-0595. Epub 2022 Aug 24. PMID 36000541